CLINICAL TRIAL: NCT03268109
Title: COGnitive ImpairmenT in Older HIV-infected Patients ≥ 65 Years Old.
Acronym: COGITO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2017_3
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Memory Impairment; HIV/AIDS; Cognitive Impairment
MeSH Terms: conditions — Memory Disorders; Acquired Immunodeficiency Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- people living with HIV: subjects infected with HIV and with cognitive complaints
  Interventions: Other: assessment of cognitive impairment
- control subjects: subjects not infected with HIV and with cognitive complaints
  Interventions: Other: assessment of cognitive impairment

INTERVENTIONS:
Other: assessment of cognitive impairment — Measure of Global Deficit Score

SUMMARY:
Despite combined antiretroviral therapy (cART), milder forms of HIV-associated neurocognitive disorders (HAND) persist in 20-50% of persons living with HIV (PLHIV). Since more PLH are at risk for HAND due to aging, the frequency of HAND in PLHIV ≥ 65 years old is important to quantify for planning early intervention to attenuate both functional and occupational disabilities due to cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Personal or familial cognitive complaints
* Individual aged ≥ 65 years old and < 81 years old
* Instrumental activities of daily living (IADL) score between 3-4
* French speaking individual
* Informed consent signed For PLHIV
* HIV infection
* Undetectable HIV viral load ≥ 1 year
* Current cluster of differentiation (CD4) cell count > 100/mm3 For controls
* negative HIV serology ≤ 6 months

Exclusion Criteria:

* Opportunistic infection < 5 years
* Contraindications to MRI

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: cART-treated PLHIV ≥65 years old having a memory complaint and virologically controlled for at least 1 year and to compare PLHIV to HIV-uninfected individuals matched for age, sex and educational level
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
cognitive impairment | baseline
  cognitive impairment frequency, defined by a z-score ≤ 1.65 in at least 2 cognitive domains

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Moulignier, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild /URC, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided